CLINICAL TRIAL: NCT04892810
Title: Immunomonitoring of Interventional Radiology Procedures in the Management of Hepatocellular Carcinoma
Acronym: PAI²HCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: Grenoble University Hospital
Record Dates: First submitted 2021-05-03; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- RFA: Patient with HCC and decision of treatment with ablation
  Interventions: Procedure: Percutaneous ablation
- MWA: Patient with HCC and decision of treatment with ablation
  Interventions: Procedure: Percutaneous ablation

INTERVENTIONS:
Procedure: Percutaneous ablation — Hepatic Percutaneous Ablation with radiofrequency or microwave

SUMMARY:
This cohort study compares immune response induced in two groups of small HCC patients treated by ablation (group1 RFA, group 2 MWA). Patients will benefit for tumoral and non tumoral biopsies prior to treatment and stepped peripheral blood samples juste before ablation and during the first month after.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven HCC for less than 3 months before ablation
* Decision of ablation treatment in multidisciplinary meeting

Exclusion Criteria:

* Fibrolamellar HCC
* Hepatocholangiocarcinoma

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 40 years old that can benefit for ablation (either RFA or MWA) for HCC
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-05-31 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
To compare induced immunomodulation by RFA and MWA in HCC patients | one month
  Comparison of modulation of immune cells (frequency, activity, function) between the two groups. Study of immune cells will include T cells with immune checkpoints molecules (PD-1+ CD8+ T, 4-1BB+ CD8+ T, LAG-3+ CD8+ T, Tim-3+ CD8+ T, COS+ CD8+ T) before and after the treatment (day 0, day 2, day 7, day 30)

SECONDARY OUTCOMES:
To evaluate early induced immunomodulation after RFA in HCC patients | one month
  Differences of frequencies, activities, functions of immune cells before and after the RFA treatment (day 0, day 2, day 7, day 30). Study of immune cells will include T cells with immune checkpoints molecules (PD-1+ CD8+ T, 4-1BB+ CD8+ T, LAG-3+ CD8+ T, Tim-3+ CD8+ T, COS+ CD8+ T)
To evaluate early induced immunomodulation after MWA in HCC patients | one month
  Differences of frequencies, activities, functions of immune cells before and after the MWA treatment (day 0, day 2, day 7, day 30). Study of immune cells will include T cells with immune checkpoints molecules (PD-1+ CD8+ T, 4-1BB+ CD8+ T, LAG-3+ CD8+ T, Tim-3+ CD8+ T, COS+ CD8+ T)